CLINICAL TRIAL: NCT04679636
Title: Effects of Heart Rate Variability Biofeedback on Promoting Autonomic Function and Decreasing Nicotine Withdrawal Symptoms and Dependence in Smoking Cessation Adults
Brief Title: Effects of HRV Biofeedback on Autonomic Function and Nicotine Withdrawal Symptoms and Dependence in Smoking Cessation Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Yu-Ju Chen, Dean of nursing, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2-2020-1204
Record Dates: First submitted 2020-12-18; First posted 2020-12-22 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Heart Rate Variability, Biofeedback, Nicotine Dependence, Nicotine Withdrawal, Anxiety, Depression, Insomnia
MeSH Terms: conditions — Tobacco Use Disorder; Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): receive biofeedback training for heart rate variability for eight weeks
  Interventions: Behavioral: heart rate variability biofeedback
- Control group (No Intervention): receive conventional treatment

INTERVENTIONS:
Behavioral: heart rate variability biofeedback — receive biofeedback training for heart rate variability for eight weeks
  Arms: Experimental group

SUMMARY:
This study is a randomized controlled trial. It is estimated that 80 quitters will be recruited, and they will be randomly included in the experimental group and 40 in the control group. The experimental group will be involved in heart rate variability biological feedback training for eight weeks, and the control group will receive conventional treatment. Use the scale to assess the symptoms of nicotine withdrawal-anxiety, depression and insomnia, as well as the degree of nicotine dependence before and after the intervention; the autonomic nervous function of the participants was measured by heart rhythm variation before and after the intervention; in addition, the cessation of smoking was tracked by telephone once a month for six Months. Discuss interventional biological feedback training and evaluate its effectiveness in improving heart rate variability, which represents autonomic nervous function, and alleviating nicotine withdrawal anxiety, insomnia, and depression symptoms, as well as nicotine dependence.

DETAILED DESCRIPTION:
Smoking cessation has been one of the priorities in public health for many years, because the severity of the disease and the social and economic losses caused by smoking cannot be ignored. Among them, nicotine dependence is one of the important issues in quitting smoking. Nicotine withdrawal symptoms often make the quitters' actions fail, especially anxiety, insomnia, and depression, which further affect the lives of quitters. If an intervention can be provided to improve the nicotine withdrawal symptoms of quitters and reduce nicotine dependence, it should be able to improve the effectiveness of smoking cessation.This study is a randomized controlled trial to facilitate sampling. It is expected that 80 quitters will be recruited at the smoking cessation clinic of the medical center through the referral of the attending physician, and 40 will be randomly included in the experimental group and the control group. The experimental group will receive biofeedback training for heart rate variability for eight weeks, while the control group will receive conventional treatment. Use the scale to assess nicotine withdrawal symptoms before and after intervention-the degree of anxiety (Beck Anxiety Inventory), depression (Beck Depression Inventory) and insomnia (Pittsburgh Sleep Quality Index), And the degree of nicotine dependence (Nicotine Dependence Scale; Fagerstrom Test for Nicotine Dependence); the autonomic nerve function of the participants was measured by heart rhythm variability before and after the intervention; in addition, the cessation of smoking was tracked by telephone once a month for six months. This study is mainly to explore interventional biological feedback training to evaluate its effectiveness in improving the representative autonomic nervous function-heart rate variability and alleviating nicotine withdrawal anxiety, insomnia and depression symptoms and nicotine dependence.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to quit smoking
2. Clear consciousness
3. Able to communicate in Mandarin or Taiwanese

Exclusion Criteria:

1. Diagnosed with asthma or chronic obstructive pulmonary disease
2. Diagnosed with nervous system
3. Diagnosis of mental illness
4. Arrhythmia, use of cardiac pacemakers, and atrioventricular conduction disorders

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-11-26 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
autonomic nerve function | baseline
  heart rate variability index
autonomic nerve function | 1 month
  heart rate variability index
autonomic nerve function | 2 month
  heart rate variability index
autonomic nerve function | 6 month
  heart rate variability index

SECONDARY OUTCOMES:
symptom distress(Anxiety) | baseline
  Beck Anxiety Inventory
symptom distress(Anxiety) | 1 month
  Beck Anxiety Inventory
symptom distress(Anxiety) | 2 month
  Beck Anxiety Inventory
symptom distress(Anxiety) | 6 month
  Beck Anxiety Inventory
symptom distress(Depression) | baseline
  Beck Depression Inventory-II
symptom distress(Depression) | 1 month
  Beck Depression Inventory-II
symptom distress(Depression) | 2 month
  Beck Depression Inventory-II
symptom distress(Depression) | 6 month
  Beck Depression Inventory-II
symptom distress(Sleep) | baseline
  Pittsburgh Sleep Quality Index
symptom distress(Sleep) | 1 month
  Pittsburgh Sleep Quality Index
symptom distress(Sleep) | 2 month
  Pittsburgh Sleep Quality Index
symptom distress(Sleep) | 6 month
  Pittsburgh Sleep Quality Index
Cigarette Dependence | baseline
  Short-Form Cigarette Dependence Questionnaire
Cigarette Dependence | 1 month
  Short-Form Cigarette Dependence Questionnaire
Cigarette Dependence | 2 month
  Short-Form Cigarette Dependence Questionnaire
Cigarette Dependence | 6 month
  Short-Form Cigarette Dependence Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service Medical Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No